CLINICAL TRIAL: NCT02266992
Title: Exploring Novel Mechanisms of Vaccine Failure and Induction of Pulmonary Immunity Following Live Attenuated Influenza Vaccination in HIV-infected Individuals: a Pilot Study.
Brief Title: Exploring Novel Mechanisms of Vaccine Failure LAIV Pilot Study
Acronym: LAIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STH18166
Record Dates: First submitted 2014-10-06; First posted 2014-10-17 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Acquired Immune Deficiency Syndrome Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluenz Tetra (Experimental): Live attenuated influenza vaccine- Fluenz tetra. Intra-nasal administration of 0.2ml (0.1ml in each nostril).
  Interventions: Biological: Live attenuated Vaccine- Fluenz Tretra

INTERVENTIONS:
Biological: Live attenuated Vaccine- Fluenz Tretra — Intra-nasal administration of 0.2ml (0.1ml in each nostril).

SUMMARY:
Influenza ('flu) can cause severe infections, especially in people with weakened immune systems such as those with HIV. For this reason, yearly vaccination is recommended with the standard 'inactivated' influenza vaccine to try and prevent infections in these populations. It is also recommended in all health care workers, to help prevent the spread of influenza within healthcare settings. However, having HIV infection may mean vaccines work less well in some people and the investigators do not completely understand why. An alternative to the standard 'inactivated' annual influenza vaccine is the 'live attenuated influenza vaccine' (LAIV), which means it consists of weakened versions of the influenza virus.

Unlike the standard vaccine, which is given by injection, LAIV is a spray that is given into each nostril. It is now given to children in the UK in preference to the standard vaccine as it results in greater protection from influenza. In some other countries, like the USA, adults are also given LAIV, where it seems to work just as well as the standard vaccine. A few studies in the past have shown that LAIV is safe and effective in HIVinfected children and adults. The investigators want to give LAIV to HIVinfected and HIV negative individuals, to try to find out new information about how HIV infection may change the way in which people respond to vaccines. The investigators will do this by comparing both the early genetic response to the vaccines and later responses from cells specifically targeted to fight influenza ('Tcells'), in these groups. In the long term, the investigators hope that this will lead to designing new ways of improving the response to vaccines in HIVinfected people. As LAIV is given into each nostril, rather than an injection, the investigators also want to see if LAIV results in Tcells in the lung that are specifically targeted to fight influenza

DETAILED DESCRIPTION:
The emerging field of systems vaccinology offers an unbiased, global approach to studying immune responses to vaccines, unlike the traditional reductionist approaches that focus on specific arms of the immune system (1,2).

Recent work has studied responses to the trivalent inactivated influenza vaccine (TIV) and intranasal live attenuated influenza vaccine (LAIV) in immunocompetent adults, showing contrasting early transcriptional signatures elicited by the two vaccines (3). LAIV induces type I interferon related genes, antigen presenting cells (3) and mucosal IgA (4), suggesting that protection may be conferred via mucosal immunity and Tcells primed by early innate responses (5,6), rather than the TIV induced systemic antibody response. This approach has revealed novel insights into how early molecular signatures (e.g. expression of Calcium/calmodulin dependent kinase IV) correlates with later humoral immune responses, but similar relationships between innate and Tcell responses in response to LAIV remain unexplored3.

Influenza is a common respiratory viral infection in HIV infected individuals worldwide, who are at a greater risk of severe infection even in the antiretroviral therapy (ART) era (7,8). Although immunization with TIV reduces these risks, as with other vaccines in HIVinfected individuals (9,10), TIV is poorly immunogenic in the immunosuppressed and new strategies are required to optimise protective immunity (1114). A systems vaccinology approach comparing the effects of LAIV in HIV infected and uninfected adults could reveal novel mechanisms of vaccine failure in those with suboptimal vaccine responses and in turn lead to potential ways of subverting this immune defect (2).

LAIV is licensed for use in healthy children and adults aged 2 - 49 years in the United States of America. It has also been introduced for vaccination of children in the UK in 2013 onwards, with a license for use in children and adolescents aged 24 months to 18 years of age (including those with asymptomatic HIV infection). Although initial concerns existed about the safety of LAIV in HIV infected individuals, several studies in both children and adults have not demonstrated any significant adverse effects (1518). A large study that administered either LAIV (n = 122) or TIV (n = 121) to HIV infected children (mean age 12) found the safety profile of the two vaccines to be similar (including incidence of pulmonary symptoms), other than an increased incidence of injection site reactions in the TIV arm (17).

No effect on CD4 count or viral load was observed. Approximately 23% of children were found to shed vaccine strains of influenza within the first week following vaccination, which is similar to rates in HIV negative children. A study of HIV infected (n = 57) and uninfected (n = 54) adults also reported a similar safety profile, with rates of reactogenicity following LAIV equivalent between the two groups, but also no different to placebo arms, other than an increase in mild self limiting rhinorrhea and nasal congestion in the LAIV arms (16). Interestingly, in contrast to studies in children, only one adult was found to shed vaccine influenza strains, which is likely due to the attenuated nature of LAIV and preexisting antiinfluenza immunity in adults. While traditionally HIV infection is a relative contraindication to live vaccine administration, there is also now good experience with safely using live vaccines such as the Yellow Fever vaccine in subjects with CD4 counts >200/mm3 (19) and is included in travel vaccination guidance for HIV infected individuals who meet these criteria (20). Recent guidance on immunisation of immunocompromised adults also recommends the use of live varicella vaccine in HIV infected adults who are not severely immunocompromised and are nonimmune to varicella (20). As live vaccines typically induce a more potent immune response than inactivated or subunit vaccines, this approach warrants further investigation in HIV infected subjects. While LAIV is more immunogenic than TIV in children (21,22), data suggests that LAIV and TIV have similar effectiveness in preventing influenza in healthy adults, despite lower antibody seroconversionin LAIV (23,24). LAIV is more likely to confer protection via innate immune priming of mucosal cellular responses (3,23,24). In addition, LAIV may provide protection against mismatched strains of influenza (21,22) and unlike TIV, result in protective immunity that extends beyond the year of administration (25).

The importance of Tcell responses in reducing the severity of influenza is increasingly recognised (26) and may be a better correlate of protection than antibodies in the elderly (2729). Murine data have demonstrated the role of LAIV elicited pulmonary influenza specific CD8+ Tcells, in providing longlived protection against subsequent viral challenge (3032), although this is yet to be confirmed in human studies. This protection appears to extend to heterologous viruses, as the Tcell response is directed primarily at internal proteins, which are conserved across many strains. This is important, given the ongoing threat of new emerging influenza viruses.

HIV infected subjects have impaired naturally acquired influenza specific Tcell responses in both blood and lung (33,34). No human studies exist on the degree of pulmonary Tcell immunity induced by LAIV in HIV infected or immunocompetent adults. No studies have also used a systems biology approach to study the immune response to live vaccine challenge in HIVinfection. While HIVinfected subjects may display an aberrant systemic immune response to LAIV, it could also provide a useful strategy to induce potent heterotypic mucosal immunity in a population who display suboptimal responses to TIV. The study will be conducted in compliance with the protocol, Good Clinical Practice (GCP) and the applicable NHS R&D Form IRAS Version 3.5 8 155866/618731/14/528 many strains. This is important, given the ongoing threat of new emerging influenza viruses.

HIV infected subjects have impaired naturally acquired influenza specific Tcell responses in both blood and lung (33,34). No human studies exist on the degree of pulmonary Tcell immunity induced by LAIV in HIV infected or immunocompetent adults. No studies have also used a systems biology approach to study the immune response to live vaccine challenge in HIV infection. While HIV infected subjects may display an aberrant systemic immune response to LAIV, it could also provide a useful strategy to induce potent heterotypic mucosal immunity in a population who display suboptimal responses to TIV. The study will be conducted in compliance with the protocol, Good Clinical Practice (GCP) and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age18 - 49
* HIV1 infected
* On antiretroviral therapy
* CD4 count of >200/mm3 (for at least 6 months, last available measurement within 3 months)
* Viral load undetectable (for at least 6 months, last available measurement within 3 months)
* Historyof having received at least one dose of trivalent inactivated influenza vaccine in the past
* Nonsmoker

Exclusion Criteria:

* Severe egg allergy
* Hypersensitivity to gentamicin
* Pregnant or breastfeeding
* Chronic lung disease (e.g. bronchiectasis)
* A history of severe asthma or current active wheezing
* Other cause for immunosuppression (e.g. malignancy) or immunosuppressive medication
* Hepatitis B or C coinfection (as defined by a detectable HBSAg or HCV RNA)
* Planned close contact with severely immunocompromised individuals in 2 weeks following LAIV (e.g bone marrow transplant recipients)
* Recipient of any other vaccination within the last 4 weeks
* Individuals who have had a febrile illness or other symptoms of acute infectious illness (respiratory, enteric or soft tissue) within the last 2 weeks.
* Individuals with a known and current history of anaemia or any symptoms (shortness of breath, chronic fatigue, chest pain or pallor) suggestive of possible anaemia or haemoglobin below the lower limit of sex adjusted normal range on a full blood count taken within the last 3 months.
* Current(active) participation in any clinical trial
* Inability to communicate in English or convey willingness to participate.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Differential gene expression at day 3 following administration of LAIV from baseline, via DNA microarrays. | day 3
  Do HIVinfected individuals have distinct differential early gene expression profiles following intranasal live attenuated influenza vaccine, when compared to age and sexmatched HIVnegative subjects, thus providing insights into the aberrant immunological response to live vaccines modulated by HIV infection?

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation trust, Sheffield, South Yorkshire, United Kingdom